CLINICAL TRIAL: NCT01554930
Title: A Clinical Trial to Evaluate the Effectiveness and Safety of Chinese Medicine in the Treatment of Severe Type of Hand, Foot, and Mouth Disease
Brief Title: Effectiveness and Safety of Chinese Medicine to Treat Hand, Foot, and Mouth Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Collaborators: China Academy of Chinese Medical Sciences (Other); Beijing YouAn Hospital (Other); The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other); Beijing University of Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200907001-3
Record Dates: First submitted 2012-03-11; First posted 2012-03-15 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Hand, Foot, and Mouth Disease
Keywords: HFMD; Traditional Chinese Medicine; Xiyanping
MeSH Terms: conditions — Hand, Foot and Mouth Disease | interventions — Mannitol; Methylprednisolone; Immunoglobulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Western therapy (Active Comparator)
  Interventions: Drug: Western therapy (mannitol, methylprednisolone, immunoglobulin, febrifuge)
- Xiyanping injection plus western therapy (Experimental)
  Interventions: Drug: Xiyanping injection plus western therapy

INTERVENTIONS:
Drug: Western therapy (mannitol, methylprednisolone, immunoglobulin, febrifuge) — Mannitol:0.5-1.0g/kg，q4h to q8h ivgtt; Methylprednisolone:1mg-2mg/kg·d,qd iv; Immunoglobulin：1g/kg; Others:febrifuge，sedative，etc.
  Arms: Western therapy
Drug: Xiyanping injection plus western therapy — Xiyanping injection:5-10mg/kg/d (0.2-0.4ml/kg/d),qd ivgtt; Mannitol:0.5-1.0g/kg，q4h to q8h ivgtt; Methylprednisolone:1mg-2mg/kg·d,qd iv; Immunoglobulin：1g/kg; Others:febrifuge，sedative，etc.
  Arms: Xiyanping injection plus western therapy

SUMMARY:
The study is aimed to evaluate the effectiveness and safety of Xiyanping injection,a traditional Chinese medicine (TCM), in the treatment of severe type of hand, foot, and mouth disease (HFMD).

DETAILED DESCRIPTION:
By adopting a multi-center, randomized and controlled clinical trial, this study is aimed to evaluate the effectiveness, safety and economic evaluation of a traditional Chinese medicine, Xiyanping injection,for treatment of HFMD, and to provide scientific evidence for the construction of TCM methods in treating HFMD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of severe hand-foot-mouth disease patients according to Hand-Foot-Mouth Disease Treatment Guidelines 2010 issued by China's Ministry of Health; More than 1/3 patients should be diagnosed by etiological examination.
* Less than 24 hours of occurrence of fever and/or occurrence of tetter or herpes.
* Age of 1-13 years.
* Patients or their guardians agree to participate in this study and signed the informed consent form.

Exclusion Criteria:

* Complicated with other diseases such as neurogenic pulmonary edema, cardiopulmonary failure.
* Complicated with other serious primary diseases in organ such as congenital heart disease, chronic hepatitis, nephritis and blood diseases, etc.
* With history of allergies on traditional Chinese medicine.
* Patients who using glucocorticoids for based diseases.
* Patients who having history of hemolysis.
* Patients or their guardians suffering from Psychiatric diseases.
* Attending other clinical studies on HFMD after diagnosed.

Ages: 1 Year to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
complication rate | 15 days
  Refering to the ratio of patient having complications such as pulmonary edema, myocarditis，damage of central nervous system，shock, respiratory failure, multiple organ failur etc.

SECONDARY OUTCOMES:
time of body temperature going back to normal | 15 days
  Refering to the time of the armpit temperature of lower than 37.0 degrees Celsius, lasting for at least 24 hours, after the medicine is taken.
time of symptom disappearance | 15 days
  Referring to the length of time when clinical symptoms and signs totally disappear after the medicine is used.
safety outcome | 15 days
  Calculated by adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Li Xiu hui, PhD, Study Chair — Beijing You-An Hospital; Zhang Guo liang, PhD, Study Chair — The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine; Shi Qin sheng, PhD, Principal Investigator — Handan Maternal and Child Health Care Hospital; Zhu Qin xiong, PhD, Principal Investigator — Jiangxi Children's Hospital; Yang tong, PhD, Principal Investigator — LiuZhou People's Hospital
Locations (3):
- China (3):
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Handan Maternal and Child Health Care Hospital, Handan, Hebei
  - Jiangxi Children's Hospital, Nanchang, Jiangxi

REFERENCES:
- [Background] Hamaguchi T, Fujisawa H, Sakai K, Okino S, Kurosaki N, Nishimura Y, Shimizu H, Yamada M. Acute encephalitis caused by intrafamilial transmission of enterovirus 71 in adult. Emerg Infect Dis. 2008 May;14(5):828-30. doi: 10.3201/eid1405.071121. PMID 18439374
- [Background] Hosoya M, Kawasaki Y, Sato M, Honzumi K, Hayashi A, Hiroshima T, Ishiko H, Kato K, Suzuki H. Genetic diversity of coxsackievirus A16 associated with hand, foot, and mouth disease epidemics in Japan from 1983 to 2003. J Clin Microbiol. 2007 Jan;45(1):112-20. doi: 10.1128/JCM.00718-06. Epub 2006 Nov 8. PMID 17093028
- [Background] Yoke-Fun C, AbuBakar S. Phylogenetic evidence for inter-typic recombination in the emergence of human enterovirus 71 subgenotypes. BMC Microbiol. 2006 Aug 30;6:74. doi: 10.1186/1471-2180-6-74. PMID 16939656
- [Background] Chang LY, King CC, Hsu KH, Ning HC, Tsao KC, Li CC, Huang YC, Shih SR, Chiou ST, Chen PY, Chang HJ, Lin TY. Risk factors of enterovirus 71 infection and associated hand, foot, and mouth disease/herpangina in children during an epidemic in Taiwan. Pediatrics. 2002 Jun;109(6):e88. doi: 10.1542/peds.109.6.e88. PMID 12042582
- [Background] Shen WC, Chiu HH, Chow KC, Tsai CH. MR imaging findings of enteroviral encephaloymelitis: an outbreak in Taiwan. AJNR Am J Neuroradiol. 1999 Nov-Dec;20(10):1889-95. PMID 10588115